CLINICAL TRIAL: NCT05020652
Title: A Randomized, Double Blind, Double Dummy, Parallel Controlled, Multicenter Phase II Clinical Trial of TQ05105 Tablets Versus Hydroxyurea Tablets in the Treatment of Moderate and High Risk Myelofibrosis
Brief Title: A Clinical Trial of TQ05105 Tablets in the Treatment of Moderate and High Risk Myelofibrosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQ05105-II-01
Record Dates: First submitted 2021-08-23; First posted 2021-08-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Moderate and High Risk Myelofibrosis
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Hydroxyurea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQ05105 tablets + Hydroxyurea blank tablets (Experimental): Take TQ05105 Tablets + Hydroxyurea blank tablets orally on an empty stomach, with an interval of at least 8 hours, and the best interval is 12 hours. Every 4 weeks is a period of administration
  Interventions: Drug: TQ05105 tablets
- TQ05105 blank tablets + Hydroxyurea tablets (Active Comparator): Take TQ05105 blank tablets + Hydroxyurea tablets orally on an empty stomach, with an interval of at least 8 hours, and the best interval is 12 hours. Every 4 weeks is a period of administration
  Interventions: Drug: Hydroxycarbamide tablets

INTERVENTIONS:
Drug: TQ05105 tablets — TQ05105 tablet is a JAK2 inhibitor, which can be used to treat JAK2 target related diseases, such as moderate or high-risk multiple myelofibrosis.
  Arms: TQ05105 tablets + Hydroxyurea blank tablets
Drug: Hydroxycarbamide tablets — Hydroxycarbamide tablet is a nucleoside diphosphate reductase inhibitor.
  Arms: TQ05105 blank tablets + Hydroxyurea tablets

SUMMARY:
Q05105 tablet is a Janus kinase 2 (JAK2) inhibitor, which can be used to treat JAK2 target related diseases, such as moderate or high-risk multiple myelofibrosis

ELIGIBILITY:
Inclusion Criteria:

1. The subjects volunteered to join the study and signed informed consent, with good compliance;
2. Age: 18-75 years old (when signing the informed consent form); Eastern Cooperative oncology Group (ECoG) Performance Status (PS) score: 0-2; The expected survival time is more than 24 weeks;
3. Primary Myelofibrosis (PMF) was diagnosed according to World Health Organization (WHO) standard (2016 Edition), or Post Polycythemia Vera(PV)-MF or Post Essential Thrombocythemia (ET)-MF was diagnosed according to International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) standard; JAK2 mutation or not was included in the study;
4. According to Dynamic International Prognostic Scoring System (DIPSS) prognosis grading criteria, the patients with myelofibrosis were assessed as medium risk (including medium risk-1, medium risk-2) or high risk;
5. Splenomegaly: palpate the splenic margin at least 5cm below the ribs (the distance from the costal margin to the farthest point of splenic protrusion);
6. Peripheral blood primordial cells ≤ 10%;
7. If antifibrotic treatment for myelofibrosis is ongoing before screening, hydroxyurea, any immunomodulators such as thalidomide, short-acting interferons, androgenic drugs, and any immunosuppressants (such as prednisone > 10mg/day or equivalent strength corticosteroids) must be discontinued for at least 2 weeks before randomization; long-acting interferons and erythropoietin must be discontinued for at least 4 weeks before randomization;
8. No growth factor, colony stimulating factor, thrombopoietin or platelet transfusion was received within 2 weeks before the examination, and hemoglobin (Hgb) ≥ 80g / L, platelet count (PLT) ≥ 100 within 7 days before the random date × 10^9 / L and neutrophil absolute value (neut) ≥ 1.0 × 10^9/L;
9. The main organs were functional 7 days before the random date, which was in accordance with the following criteria: Total Bilirubin (TBIL) was less than 2 times the upper limit of normal value (ULN); Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) were less than 2.5 times of ULN; Serum creatinine (Cr) < 1.5 times of ULN or creatinine clearance rate (Ccr) ≥ 50ml/min; The blood coagulation function should be checked in accordance with: prothrombin time (PT), activated partial thromboplastin time (APTT), international standardized ratio (INR) < 1.5 × ULN (not anticoagulant treatment); Left ventricular ejection fraction (LVEF) evaluated by color Doppler ultrasonography ≥ 50%;
10. Female subjects of childbearing age should agree to use contraceptive measures (such as intrauterine device, contraceptive or condom) during the study period and within 6 months after the end of the study; The serum pregnancy test was negative within 7 days before the date of randomization and must be non lactating subjects; Male subjects should agree to use contraception during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

1. Those who have received allogeneic stem cell transplantation in the past, or autologous stem cell transplantation within 3 months before the random date, or recently planned stem cell transplantation;
2. Patients who have received JAK inhibitors in the past;
3. Those who had undergone splenectomy or received splenic radiotherapy within 6 months before the date of randomization (including internal and external radiotherapy);
4. Other malignancies were present or present within 3 years before the date of randomization. The following two cases can be included: other malignant tumors treated by single operation have achieved 5-year disease-free survival (DFS) in a row; Cured cervical carcinoma in situ, non melanoma skin cancer and superficial bladder tumor [ta (non-invasive tumor), tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];
5. Patients with multiple factors (such as inability to swallow, postoperative gastrointestinal resection, acute and chronic diarrhea, intestinal obstruction, etc.) affecting oral or absorption of drugs;
6. Non hematological toxicity caused by previous treatment did not return to ≤ 1 (excluding alopecia);
7. Patients who received major surgical treatment or had obvious traumatic injury within 4 weeks before the date of randomization;
8. At present, there are congenital bleeding or coagulation diseases, or are using anticoagulant therapy;
9. Arteriovenous thrombotic events occurred within 6 months before the random date, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism;
10. A history of psychotropic substance abuse or mental disorder;
11. Active or uncontrolled severe infection (≥ Common Terminology Criteria for Adverse Events(CTCAE)2 infection);
12. Hepatitis B Virus (HBV) DNA≥ULN； Hepatitis C antibody positive and Hepatitis C Virus (HCV) RNA ≥ ULN;
13. Myocardial ischemia or myocardial infarction, arrhythmia, QT interval prolongation (corrected QT interval (QTc) ≥ 450 ms for male, QTc ≥ 470 ms for female) and congestive heart failure (NYHA classification) of grade 2 or above;
14. Blood pressure control is not ideal (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg);
15. Renal failure requires hemodialysis or peritoneal dialysis;
16. Newly diagnosed pulmonary fibrosis or drug-related interstitial lung disease within 3 months before the date of randomization;
17. History of immunodeficiency, including Human Immunodeficiency Virus (HIV) positive or other acquired or congenital immunodeficiency diseases, or organ transplantation;
18. Patients with epilepsy and need treatment;
19. Within 4 weeks prior to the random date, the patient had received chemotherapy, radiotherapy or other anti-cancer treatments (except as stipulated in item 7 of the inclusion criteria);
20. Within 2 weeks before the date of randomization, he received Chinese patent medicines (including compound cantharis capsule, Kang'ai injection, kang'laite capsule / injection, Aidi injection, Brucea javanica oil injection / capsule, Xiaoaiping tablet / injection, cinobufagin capsule, etc.) with anti-tumor indications specified in nmpa approved drug instructions;
21. Uncontrolled pleural effusion, pericardial effusion or ascites;
22. Patients with central nervous system involvement;
23. There was a history of live attenuated vaccine inoculation within 4 weeks before the date of randomization or live attenuated vaccine inoculation was planned during the study period;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Spleen Volume was Reduced by more than 35% from baseline（SVR35） assessed by Independent Review Committee (IRC) | up to 24 weeks
  Proportion of subjects whose spleen volume was reduced by more than 35% from baseline at the end of week 24 of IRC assessment (SVR35)

SECONDARY OUTCOMES:
SVR35 assessed by the researchers and objective response rate (ORR) | up to 24 weeks
  Proportion of subjects whose spleen volume was reduced by more than 35% from baseline to the end of the 24th week assessed by the researchers and ORR
optimal response rate of splenic response | up to 120 weeks
  Proportion of subjects with at least one reduction in spleen volume ≥ 35% from baseline.
onset time of splenic response | up to 120 weeks
  The time between the date of randomization and the date when the spleen volume decreased ≥ 35% from the baseline for the first time.
Duration of Maintenance of a Least 35% Reduction in Spleen Volume(DoMSR) | up to 120 weeks
  Duration of spleen volume reduction ≥ 35% from baseline (domsr): the time between the date when the spleen volume reduction ≥ 35% from baseline occurs for the first time and the date when the spleen volume reduction < 35% from baseline.
the proportion of subjects whose total symptom score of Myeloproliferative neoplasm- Symptom Assessment Form- Total Symptom Score(MPN-SAF TSS) decreased by more than 50% compared with baseline | up to 24 weeks
  At the 24th week, the proportion of subjects whose total symptom score of MPN-SAF TSS) decreased by more than 50% compared with baseline.
The total symptom score of MPN-SAF TSS decreased compared with baseline | up to 24 weeks
  The total symptom score of MPN-SAF TSS decreased compared with baseline;
Progression-free survival (PFS) | up to 120 weeks
  The interval from the random date to the date of occurrence of any of the following events, whichever occurs first: ① the spleen volume increases by ≥ 25% compared with the lowest value during the treatment period (including the screening period); ② Death from any cause; ③ Start other anti-MF treatments;
Leukemia free survival (LFS) | up to 120 weeks
  The time interval between the random date and the date of any of the following events, whichever occurs first, shall prevail: ① the date when the first bone marrow smear showed that the number of primordial cells was more than or equal to 20%; ② The first peripheral blood smear showed that the number of primordial cells was more than or equal to 20% and the absolute value of primordial cells was more than or equal to 1% × 10^9 / L for at least 2 weeks; ③ Death from any cause;
Overall survival (OS) | up to 120 weeks
  The time interval between the random date and death from any cause
The incidence and severity of adverse events (AEs) occurred during the study | up to 120 weeks
  The incidence and severity of AEs occurred during the study

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - West China School of Medicine / West China Hospital, Sichuan University, Chengdu, Sichuan
  - Institute of Hematology & Blood Diseases Hostpital, Chinese Academy of medical sciences & Peking Union Medical College, Tianjin, Tianjin Municipality